CLINICAL TRIAL: NCT02725580
Title: Phase I/IIa Gene Transfer Clinical Trial for Variant Late Infantile Neuronal Ceroid Lipofuscinosis, Delivering the CLN6 Gene by Self-Complementary AAV9
Brief Title: Gene Therapy For Children With Variant Late Infantile Neuronal Ceroid Lipofuscinosis 6 (vLINCL6) Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emily de los Reyes (Other)
Responsible Party: Sponsor-Investigator, Emily de los Reyes, Dr. Emily De Los Reyes, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-GTX-501-01
Record Dates: First submitted 2016-03-16; First posted 2016-04-01 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Variant Late-Infantile Neuronal Ceroid Lipofuscinosis
Keywords: Neuronal ceroid lipofuscinosis (NCL); CLN6; vLINCL6; Gene Transfer; CLN6 Batten Disease; Batten Disease
MeSH Terms: conditions — Ceroid Lipofuscinosis, Neuronal, 6; Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Participants with diagnosis of vLINCL6 Batten disease will receive a single intrathecal injection of AT-GTX-501 into the lumbar spinal cord region.
  Interventions: Genetic: AT-GTX-501

INTERVENTIONS:
Genetic: AT-GTX-501 — CLN6 Gene delivered by Self-Complementary AAV9
  Other Names: scAAV9.CB.CLN6

SUMMARY:
This is a phase 1/2, open-label, single dose study to evaluate the safety and efficacy of AT-GTX-501 delivered intrathecally into the lumbar spinal cord region of participants with mild to moderate variant late infantile neuronal ceroid lipofuscinosis associated with mutation(s) in the CLN6 gene (vLINCL6 disease).

DETAILED DESCRIPTION:
This is an open-label, single-dose study of AT-GTX-501 administered by a single intrathecal injection. Safety and efficacy are evaluated over a 2 year period. The efficacy assessments in this study are to evaluate motor, language, visual, and cognitive function, as well as survival and other outcome measures. Participants are tested at baseline, receive AT-GTX-501 on Day 0, and return for visits on Days 7, 14, 21, and 30, and then every 3 months until Month 24. Following completion of this study, there is a long-term follow up study in which data will continue to be collected (Study AT-GTX-501-02 / NCT04273243).

For more information about this study, please contact Amicus Therapeutics Patient Advocacy at clinicaltrials@amicusrx.com or +1 609-662-2000.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of vLINCL6 disease determined by genotype available at screening
2. A score of ≥ 3 on the quantitative clinical assessment of the Hamburg motor-language aggregate scale at screening
3. Aged ≥ 1 year
4. Ambulatory or able to walk with assistance

Exclusion Criteria:

1. Presence of another inherited neurologic disease, for example, other forms of Batten disease (also known as NCL) or seizures unrelated to vLINCL6 disease (participants with febrile seizures may be eligible at discretion of the investigator.)
2. Presence of another neurological illness that may have caused cognitive decline (for example, trauma, meningitis, hemorrhage) before screening
3. Active viral infection (includes human immunodeficiency virus or serology positive for hepatitis B or C)
4. Has received stem cell or bone marrow transplantation for vLINCL6 disease
5. Contraindications for intrathecal administration of the product or lumbar puncture, such as bleeding disorders or other medical conditions (for example, spina bifida, meningitis, or clotting abnormalities)
6. Contraindications for magnetic resonance imaging scans (for example, cardiac pacemaker, metal fragment or chip in the eye, aneurysm clip in the brain)
7. Episode of generalized motor status epilepticus within 4 weeks before the gene transfer visit (Visit 2)
8. Severe infection (for example, pneumonia, pyelonephritis, or meningitis) within 4 weeks before the gene transfer visit (Visit 2) (Enrollment may be postponed.)
9. Has received any investigational medication within 30 days before the gene transfer visit (Visit 2)
10. Anti-AAV9 antibody titers > 1:50 as determined by enzyme-linked immunosorbent assay
11. Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the participant's ability to comply with the protocol-required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability
12. Pregnancy any time during the study (Any female participant judged by the investigator to be of childbearing potential will be tested for pregnancy.)
13. Abnormal laboratory values from screening considered clinically significant (gamma glutamyl transferase > 3 times the upper limit of normal, bilirubin ≥ 3.0 mg/dL, creatinine ≥ 1.8 mg/dL, hemoglobin < 8 or > 18 g/dL, white blood cells > 15,000 per cmm)
14. Family does not want to disclose participant's study participation with primary care physician and other medical providers.
15. History of or current chemotherapy, radiotherapy, or other immunosuppression therapy within the 30 days preceding screening (Corticosteroid treatment may be permitted at the discretion of the investigator.)
16. Has 2 consecutive abnormal liver tests at screening (> 2 times the upper limit of normal). Liver enzymes will be re-tested once if abnormal upon initial screening.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2024-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily de los Reyes, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hosptial, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AT-GTX-501: Participants received a single intrathecal injection of AT-GTX-501 into the lumbar spinal cord region.
Period: Overall Study
Arm/Group | AT-GTX-501
Started | 13
Received at Least 1 Dose of Study Drug | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who were treated with AT-GTX-501.
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: months] | 54.6 (17.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 9
  Multiple | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence And Severity Of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product, biologic, or medical device (medicinal products). An SAE is an AE occurring during any study phase (for example, baseline, treatment, or follow-up) that fulfils any of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongs existing hospitalization; results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; and results in a congenital anomaly/birth defect. All AEs that occurred after receipt of AT-GTX-501 are classified as TEAEs. A summary of serious and all other non-SAEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Up to 38.7 months
Population: Safety population: all participants who were treated with AT-GTX-501.
Measure: Count of Participants; unit: Participants
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
Participants
  Participants with TEAEs | 13
  Participants with Grade 3 (Severe) or 4 (Life-threatening) TEAEs | 5
  Participants with SAEs | 7
  Participants with TESAEs | 7

2. Secondary Outcome: Change From Baseline In Hamburg Motor And Language Scores at Month 24
Description: The Hamburg scale is an established tool to capture the rate of decline or regression. This tool was developed to document by rating motor, language, and visual functions in participants with late infantile neuronal ceroid lipofuscinosis type 2 (CLN2) Batten disease, and to collect their incidence of grand mal seizures. To assess disease progression and evaluate efficacy, the combined score of the motor and language domains of the Hamburg scale was used. Each domain was scored from 0 (no function) to 3 (normal function) for a maximal possible score of 6 for the combined score, referred to as the Hamburg Motor + Language aggregate score. The rate of decline in Hamburg Motor + Language aggregate, Motor, and Language scores were summarized using descriptive statistics.
Time Frame: Screening (Day -30 up to -2) up to Month 24
Population: Full Analysis Set (FAS): participants who were treated with AT-GTX-501 and had an analyzable outcome (Hamburg Motor + Language aggregate score) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
score on a scale
  Motor | 0.71 (0.576)
  Language | 0.32 (0.745)
  Motor + Language Aggregate | 1.03 (1.138)

3. Secondary Outcome: Change From Baseline In Unified Batten Disease Rating Scale (UBDRS) Scores At Month 24
Description: The Unified Batten Disease Rating Scale (UBDRS) was developed to monitor rate of progression. This scale includes assessment of extrapyramidal movement abnormalities and seizures, behavioral and capability assessments (Actual Vision), as well as history relevant to variant late infantile neuronal ceroid lipofuscinosis associated with mutation(s) in the CLN6 gene (vLINCL6) disease and scoring for global impression of symptom severity. A higher UBDRS subscale score indicated greater physical impairment, with zero indicating a better outcome. Subscales included Physical Assessment (range 0-84), Seizure Assessment (range 0-54), Behavioral Assessment (range 0-55) and Capability Assessment of Actual Vision and Normal Vision (range 0-14). A positive change from baseline score indicates increased impairment and a negative score indicates decreased impairment.
Time Frame: Screening (Day -30 up to -2) and Day 30 up to Month 24
Population: Full Analysis Set (FAS): participants who were treated with AT-GTX-501 and had an analyzable outcome (Unified Batten Disease Rating Scale [UBDRS]) scores at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
score on a scale
  Physical Assessment | 16.77 (13.953)
  Seizure Assessment | 2.2 (4.49)
  Behavioral Assessment | -0.4 (3.95)
  Capability Assuming Normal Vision | -1.2 (3.96)
  Capability with Actual Vision | -0.8 (4.22)

4. Secondary Outcome: Change From Baseline In Mullen (Age-Equivalent) Scales Of Early Learning At Month 24
Description: The Mullen Scales of Early Learning were utilized to assess cognitive and motor ability in 4 areas (visual reception, fine motor, expressive language, and receptive language) in infants and children. Raw scores range from 0-50 for visual reception, 0-49 for fine motor, 0-50 for expressive language, and 0-48 for receptive language. Lower scores from baseline indicated increased developmental delay and higher scores from baseline indicated decreased developmental delay. A positive change from baseline score indicates decreased developmental delay and a negative score indicates increased developmental delay.
Time Frame: Screening (Day -30 up to -2) and Month 24
Population: Full Analysis Set (FAS): participants who were treated with AT-GTX-501 and had an analyzable outcome (Mullen [Age-Equivalent] Scales Of Early Learning score) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
score on a scale
  Visual Reception | -9.8 (10.94)
  Fine Motor | -6.8 (6.27)
  Receptive Language | -9.9 (10.69)
  Expressive Language | -7.2 (10.74)

5. Secondary Outcome: Change From Baseline In Preschool Language Scales-5th Edition (PLS-5) (Age-Equivalent) At Month 24
Description: The Preschool Language Scales-5th Edition (PLS-5) (Age-Equivalent) was a comprehensive developmental language assessment. Standard scores from each domain (auditory comprehension, expressive communication, and total language) range from 50-150. Standard scores between 85 and 115 are considered to be within normal limits. Total scores are the sum of standard scores for auditory comprehension and expressive communication, which is then converted to a total standard score using PLS-5 Appendix B. Age-equivalent scores in each area were summarized by study visit with descriptive statistics. Higher scores represent better language development and lower scores reflect a possible language delay or disorder. A positive change from baseline score indicates better language development.
Time Frame: Screening (Day -30 up to -2) and Month 24
Population: Full Analysis Set (FAS): participants who were treated with AT-GTX-501 and had an analyzable outcome (Preschool Language Scales-5th Edition [PLS-5] [Age-Equivalent] scores) at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 13
score on a scale
  Auditory Comprehension | -7.8 (12.02)
  Expressive Communication | -3.9 (10.21)
  Total Language Score | -5.7 (11.61)

6. Secondary Outcome: Change From Baseline In Development Profile-3 At Month 24
Description: The Development Profile-3 was used to screen for developmental delays in 5 areas (physical [score range 0-35], adaptive behavior [0-37], social-emotional [0-36], cognitive [0-38], communication [0-34]), where lower scores indicated increased developmental delay. The General Development Score is obtained by adding the sum of standard scores for the five scales together (range 0-180). Standard Score ranges are <70 Delayed, 70-84 Below Average, 85-115 Average, 116-130 Above Average, and >130 Well Above Average. A positive change from baseline score indicates decreased developmental delay and a negative score indicates increased developmental delay.
Time Frame: Screening (Day -30 up to -2) and Month 24
Population: Full Analysis Set (FAS): participants who were treated with AT-GTX-501 and had an analyzable outcome (Development Profile-3 Score) at baseline and had scores available at Month 24.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AT-GTX-501
Number analyzed (Participants) | 2
score on a scale
  Physical: number analyzed (Participants) | 1
  Physical | -18.0 (NA) — Not estimable as only a single participant had data available at Month 24.
  Adaptive Behavior: number analyzed (Participants) | 1
  Adaptive Behavior | -42.0 (NA) — Not estimable as only a single participant had data available at Month 24.
  Social-Emotional | -38.5 (14.85)
  Cognitive | -31.0 (11.31)
  Communication | -19.5 (17.68)
  General Development: number analyzed (Participants) | 1
  General Development | -32.0 (NA) — Not estimable as only a single participant had data available at Month 24.

ADVERSE EVENTS:
Time Frame: Up to 38.7 months
Description: Safety population: all participants who were treated with AT-GTX-501.
Arm/Group | AT-GTX-501
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AT-GTX-501 (N=13)
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Myoclonic epilepsy (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AT-GTX-501 (N=13)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Precocious puberty (Endocrine disorders) | 1
Astigmatism (Eye disorders) | 1
Gaze palsy (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Fatigue (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 9
Viral infection (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastrointestinal viral infection (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Pyuria (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 4
Myoclonic epilepsy (Nervous system disorders) | 3
Atonic seizures (Nervous system disorders) | 2
Dyskinesia (Nervous system disorders) | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 2
Myoclonus (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Drooling (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Petit mal epilepsy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 4
Abnormal behaviour (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Staring (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Glycosuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Sterile pyuria (Renal and urinary disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1
Pallor (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to the nature of the disease, coupled with the impact of a global pandemic, adjustments were made to the study design to prioritize collection of primary safety and efficacy data, including development assessments through remote telehealth visits. The results of this data are presented in this posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02725580/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02725580/SAP_001.pdf